CLINICAL TRIAL: NCT02056951
Title: Interprofessional Biopsychosocial Rehabilitation to Optimize Inpatient Multidisciplinary Orthopedic Rehabilitation for Chronic Low Back Pain
Brief Title: Interprofessional Rehabilitation for Adults With Chronic Non-specific Low Back Pain
Acronym: PASTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: Deutsche Rentenversicherung (Other); University of Wuerzburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Klaus Pfeifer, Prof. Dr., University of Erlangen-Nürnberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0421-FSCP-0529
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Low Back Pain
Keywords: Rehabilitation; Treatment Outcome; Interprofessional Relations; Interdisciplinary Communication; Behavioural Exercise Therapy; Cognitive Therapy; Health Education; Workplace related information; Multicenter Study
MeSH Terms: conditions — Low Back Pain; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multidisciplinary rehabilitation (Active Comparator): The central objective of inpatient multidisciplinary orthopedic rehabilitation (MOR) is to improve functional health with the main focus on restoring and improving work ability. A MOR lasts on average 23 days with a total extent of therapy of 48 hours on average. MOR is provided by a multiprofessional team consisting of physicians, psychologists, sport therapists, physiotherapists, occupational therapists, masseurs, social workers, dieticians and nurses. The interventions are carried out mainly in open groups.
  Interventions: Procedure: Multidisciplinary rehabilitation
- Interprofessional rehabilitation (Experimental): The central objective of the interprofessional rehabilitation (PASTOR) is the development of active self-management of chronic non-specific low back pain. PASTOR is matched to the MOR with respect to the total duration and total extent of therapy, the included professions and the interventions dimensions (physical, psychological). The differences between PASTOR and MOR are characterized by, a) an integrative combination of profession related modules within a comprehensive and consistent treatment approach, b) an interprofessional and collaborative teamwork based on profession related modules, c) the use of standardized methods, media and materials by all professions in the therapeutic team d) a highly structured and detailed manual for the entire treatment process. The interventions are carried in fixed groups with eight to twelve participants.
  Interventions: Procedure: Interprofessional rehabilitation

INTERVENTIONS:
Procedure: Multidisciplinary rehabilitation — Multidisciplinary rehabilitation includes interventions from the physical and psychological dimensions:
  * health education
  * exercise therapy
  * back school
  * physical treatments
  * psychological interventions in groups and individual counselling
  * rehabilitation/social counselling.
  Arms: Multidisciplinary rehabilitation
Procedure: Interprofessional rehabilitation — Interprofessional rehabilitation includes also interventions from the physical and psychological dimensions:
  * education about low back pain
  * behavioural exercise therapy
  * coping with pain
  * relaxation
  * work related informations
  Arms: Interprofessional rehabilitation

SUMMARY:
The primary aim of the study is to analyse the long-term effectiveness of an interprofessional and interdisciplinary rehabilitation program named "PASTOR", with a biopsychosocial approach for participants with chronic non-specific low back pain (CLBP) compared to the standard inpatient multidisciplinary orthopaedic rehabilitation (MOR) in Germany. The investigators hypothesize that in adults with CLBP the rehabilitation program PASTOR would result in a significantly higher increase in functional ability 12 months after completion of the program in comparison to the standard inpatient MOR. The investigators further hypothesize that PASTOR would lead to significantly larger improvements regarding pain-related cognitions, pain coping strategies, physical activity, health-related quality of life, and back pain episodes compared to the standard inpatient MOR.

ELIGIBILITY:
Inclusion Criteria:

* M51.2 Other specified intervertebral disc displacement
* M51.3 Other specified intervertebral disc degeneration
* M51.4 Schmorl's nodes
* M51.8 Other specified intervertebral disc disorders
* M51.9 Intervertebral disc disorder, unspecified
* M53.8 Other specified dorsopathies
* M53.9 dorsopathy, unspecified
* M54.4 Lumbago with sciatica
* M54.5 Low back pain
* M54.6 Pain in thoracic spine
* M54.8 Other dorsalgia
* M54.9 Dorsalgia, unspecified

Exclusion Criteria:

* age below 18 years or over 65 years
* specific underlying diagnosis of back pain (e. g. radicular symptoms, myelopathy)
* considerably reduced health status (e.g. comorbidity)
* considerably reduced sight and hearing (not corrected)
* severe psychiatric condition as secondary diagnosis
* inability to speak German
* current application for early retirement or invalidity pension (§51 SG V - german law)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Hannover Functional Ability Questionnaire (FFbH-R) at 12 months | baseline, one year
  The FFbH-R consists of twelve items with a three-stage answering scale (2=yes; 1=yes, but with difficulty; 0=no, or only with assistance). The summary score describes the low back pain associated functional ability in activities of daily living (e.g. "Can you wash and dry yourself from head to toe?") in adults on a scale of 0% (minimum functional ability) to 100% (maximum functional ability).
  Kohlmann Th & Raspe H (1996). Der Funktionsfragebogen Hannover zur alltagsnahen Diagnostik der Funktionsbeeinträchtigung durch Rückenschmerzen (FFbH-R). Die Rehabilitation, 34, I-VIII.

SECONDARY OUTCOMES:
Health-related Quality of Life (SF-12) | baseline, three weeks, one year
  To assess mental and physical health status during the past four weeks.
  Bullinger M & Kirchberger I (1998). SF-36, Fragebogen zum Gesundheitszustand. Göttingen: Hogrefe.
Numerical rating scale (NRS) | baseline, three weeks, one year
  Three items to assess the pain intensity reported by participants at the moment, as well as during the last six months (mean and maximum pain).
  Nagel B, Gerbershagen HU, Lindena G & Pfingsten M (2002). Entwicklung und empirische Überprüfung des Deutschen Schmerzfragebogens der DGSS. Schmerz, 16 (4), 263-270.
Freiburg Questionnaire of physical activity (FFkA) | baseline, one year
  The FQPA measures the amount of physical activity in different contexts performed by the participants: occupational setting (rating: intensive movement, moderate movement, mostly sitting) as well as leisure time physical activity (e.g. gardening, stair-climbing, habitual walking and cycling, sports). It consists of eight items.
  Frey I, Berg A, Grathwohl D & Keul J (1999). Freiburger Fragebogen zur körperlichen Aktivität - Entwicklung, Prüfung und Anwendung. Sozial- und Präventivmedizin, 44, 55-64.
Pain Management Questionnaire (FESV) | baseline, three weeks, one year
  Questionnaire to assess cognitive and behavioral pain coping strategies.
  Geissner E (2001). Fragebogen zur Erfassung der Schmerzverarbeitung (FESV). Manual. Göttingen: Hogrefe.
Avoidance-Endurance Questionnaire (AEQ) | baseline, three weeks, one year
  Questionnaire to assess fear-avoidance response pattern and avoidance-endurance response pattern to pain.
  Hasenbring MI, Hallner D & Rusu AC (2009). Fear-avoidance- and endurance-related responses to pain: development and validation of the Avoidance-Endurance Questionnaire (AEQ). Eur J Pain, 13 (6), 620-628.
Change from Baseline in Hannover Functional Ability Questionnaire (FFbH-R) at 3 weeks | baseline, three weeks
  The FFbH-R consists of twelve items with a three-stage answering scale (2=yes; 1=yes, but with difficulty; 0=no, or only with assistance). The summary score describes the low back pain associated functional ability in activities of daily living (e.g. "Can you wash and dry yourself from head to toe?") in adults on a scale of 0% (minimum functional ability) to 100% (maximum functional ability).
  Kohlmann Th & Raspe H (1996). Der Funktionsfragebogen Hannover zur alltagsnahen Diagnostik der Funktionsbeeinträchtigung durch Rückenschmerzen (FFbH-R). Die Rehabilitation, 34, I-VIII.

OTHER OUTCOMES:
Tampa Scale of Kinesiophobia | baseline, three weeks, one year
  A 17-item self report checklist using a 4-point Likert scale to assess fear of movement/ re-injury.
  Vlaeyen JWS, Kole-Snijders AMJ, Boeren RGB, & Van Eek H (1995). Fear of movement/(re) injury in chronic low back pain and its relation to behavioral performance. Pain, 62(3), 363-372.
  Nigbur K, Rusu A, Hallner D & Hasenbring M (2009). Fear of movement/(re)injury in chronic pain: Preliminary validation of a German version of the Tampa Scale for Kinesiophobia. Poster presented at Pain in Europe - 6th Congress of the European Federation of IASP® Chapters (EFIC), Lisbon 2009.
Patient Health Questionnaire (PHQ) | baseline, three weeks, one year
  Löwe B, Spitzer RL, Zipfel S & Herzog W (2002). Gesundheitsfragebogen für Patienten (PHQ-D). Manual und Testunterlagen (2. Aufl.). Karlsruhe: Pfizer.
Pain Catastrophizing Scale (PCS) | baseline, three weeks, one year
  Meyer K, Sprott H & Mannion AF (2008). Cross-cultural adaptation, reliability, and validity of the German version of the Pain Catastrophizing Scale. J Psychosom Res, 64 (5), 469-478.
Self-control inventory (SSI-L) | baseline, one year
  Fröhlich S & Kuhl J (2003). Das Selbststeuerungsinventar: Dekomponierung volitionaler Funktionen. In: J. Stiensmeier-Pelster & F. Rheinberg (Hrsg.), Diagnostik von Motivation und Selbstkonzept (S. 221-258). Göttingen [u.a.]: Hogrefe.
HAPA variables | baseline, three weeks, one year
  HAPA variables include sets of items about the risk perception, self-efficacy, outcome expectations, intention, action and coping planning, and action control regarding physical activity.
  Sniehotta FF, Scholz U & Schwarzer R (2005). Bridging the intention-behaviour gap: Planning, self-efficacy, and action control in the adoption and maintenance of physical exercise. Psychol Health, 20 (2), 143-160.
  Sniehotta FF, Schwarzer R, Scholz U & Schüz B. (2005). Action planning and coping planning for long-term lifestyle change: Theory and assessment. Eur J Soc Psychol (35), 565-576.
Stage of behavior change | baseline, one year
  Stage assessment of behaviour change contains the question: Have you performed moderate physical for 30 minutes or longer on a minimum of 3 days per week? (rating: No, and I don't intend to do so - No, but I am currently thinking about that - No, but I strongly intend to do so - Yes, but it is difficult to me - Yes and it is easy to me), and a validation item ("Since when are you regularly active as you are now?")
  Lippke S, Ziegelmann J, Schwarzer R & Velicer W (2009). Validity of stage assessment in the adoption and maintenance of physical activity and fruit and vegetable consumption. Health Psychology (28), 183-193.
Graded Chronic Pain Status (GCPS) | baseline, one year
  Six items to assess the number of days with pain during the last six months, the history of pain and the functional disability due to pain (adapted for 6 months).
  Korff M von, Ormel J, Keefe FJ & Dworkin SF (1992). Grading the severity of chronic pain. Pain, 50 (2), 133-149.
Time off work for back pain | baseline, one year
  Self-reported day of sick leave due to low back pain during the last six month
Health care utilization due to low back pain | baseline, one year
  Self-reported health care utilization due to low back pain during the last six months
Job satisfaction | baseline, one year
  A 8-item self report checklist of the IRES using a 5-point Likert scale to assess job satisfaction (ranging from 1="complete agreement" to 5="complete disagreement".
  Bührlen B, Gerdes N & Jäckel WH (2005). Entwicklung und psychometrische Testung eines Patientenfragebogens für die medizinische Rehabilitation (IRES-3). Rehabilitation, 44, 63-74.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Pfeifer, Prof. Dr., Study Chair — Friedrich-Alexander-University Erlangen-Nürnberg, Institute of Sport Science and Sport
Locations (4):
- Germany (4):
  - Frankenklinik, Bad Kissingen, Bavaria
  - Klinik Franken, Reha-Zentrum Bad Steben, Bad Steben, Bavaria
  - Asklepios Klinik Schaufling, Schaufling, Bavaria
  - University of Würzburg, Department of Medical Psychology, Medical Sociology, and Rehabilitation Sciences, Würzburg, Bavaria

REFERENCES:
- [Result] Semrau J, Hentschke C, Buchmann J, Meng K, Vogel H, Faller H, Bork H, Pfeifer K. Long-term effects of interprofessional biopsychosocial rehabilitation for adults with chronic non-specific low back pain: a multicentre, quasi-experimental study. PLoS One. 2015 Mar 13;10(3):e0118609. doi: 10.1371/journal.pone.0118609. eCollection 2015. PMID 25768735
- See also: Homepage: Research funding for care-oriented research "Chronic diseases and patient orientation" — http://www.forschung-patientenorientierung.de/index.php/projects/first-funding-phase/module-two-phase-1/pastor-pfeifer.html